CLINICAL TRIAL: NCT05103046
Title: A Phase 1, First in Human, Dose-Escalation Study of UCT-03-008 in Participants With Advanced Solid Tumors
Brief Title: First in Human Study of UCT-03-008 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 1200 Pharma, LLC (Industry)
Collaborators: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCT03008-001
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Finding as Monotherapy - Part 1 (Experimental): UCT-03-008 Dose Finding
  Interventions: Drug: UCT-03-008
- Expansion as Monotherapy - Part 2 (Experimental): UCT-03-008 RP2D Expansion
  Interventions: Drug: UCT-03-008

INTERVENTIONS:
Drug: UCT-03-008 — Orally available kinase inhibitor

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of UCT-03-008 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Measurable disease, per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function

Exclusion Criteria:

* Has not recovered [recovery is defined as NCI CTCAE, version 5.0, grade ≤1] from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements
* Received prior chemotherapeutic, investigational, or other therapies for the treatment of cancer within 14 days with small molecule and within 28 days with biologic before the first dose of UCT-03-008
* Progressive or symptomatic brain metastases
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection
* History of significant cardiac disease
* History or current evidence/risk of retinopathy
* History of myelodysplastic syndrome (MDS) or AML
* History of another cancer within 3 years before Day 1 of study treatment, with the exception of basal or squamous cell carcinoma of the skin that has been definitively treated. A history of other malignancies with a low risk of recurrence, including appropriately treated ductal carcinoma in situ (DCIS) of the breast and prostate cancer with a Gleason score less than or equal to 6, are also not excluded
* If female, is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum Tolerated Dose (MTD) | 28 Days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data

SECONDARY OUTCOMES:
Maximum Plasma UCT-03-008 Concentration following single dose (Cmax) | Cycle 0(each cycle is 28 days)
  PK assessment for UCT-03-008
Maximum Plasma UCT-03-008 Concentration at steady state (Cmax,ss) | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-03-008
Minimum Plasma UCT-03-008 Concentration following single dose (Cmin) | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-003-008
Minimum Plasma UCT-03-008 Concentration at steady state (Cmin,ss) | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-003-008
Time of Maximum Plasma UCT-03-008 Concentration following single dose (Tmax) | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-03-008
Time of Maximum Plasma UCT-03-008 Concentration at steady state (Tmax,ss) | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-03-008
Area Under the Plasma Concentration-Time Curve Over Dosing Interval (AUCtau) of UCT-03-008 | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-03-008
Area Under the Plasma Concentration-Time Curve from the time of dosing to the last measurable concentration (AUClast) of UCT-03-008 | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-03-008
Apparent Clearance (CL/F) of UCT-03-008 | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-03-008
Apparent Volume of Distribution (Vz/F) of UCT-03-008 | Cycle 0 (each cycle is 28 days)
  PK assessment for UCT-03-008
Terminal Half-life (t1/2) of plasma UCT-03-008 | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-03-008
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1
Time to Response (TTR) | up to 2 years
  Time from start of treatment to complete response or partial response
Duration of Response (DOR) | up to 2 years
  Time from complete response or partial response to objective disease progression or death due to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
1 Year Overall Survival (1YOS) | 1 year
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Alex Garcia, Study Director — TRIO-US
Locations (5):
- United States (5):
  - UCLA - JCCC Clinical Research Unit, Los Angeles, California
  - Torrance Memorial, Torrance, California
  - Winship Institute of Emory University, Atlanta, Georgia
  - Mary Crowley Cancer Research, Dallas, Texas
  - START (South Texas Accelerated Research Therapeutics), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No